CLINICAL TRIAL: NCT05412121
Title: Feasibility and Acceptability of Acupressure in Patients With Rheumatoid Arthritis
Brief Title: Acupressure in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anne Murphy, House Officer, Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00206002
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Acupressure; AcuWand; MeTime
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Acupressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Acupressure (Experimental): The self-acupressure intervention will be delivered using the modified MeTime Acupressure mobile application (App) in addition to in-person or virtual instruction via study staff.
  Interventions: Device: Acupressure

INTERVENTIONS:
Device: Acupressure — The MeTime Acupressure app will be loaded onto computer tablets or smart phones by the participants. Participants will also receive an AcuWand to be used in association with the acupressure app to help participants apply the correct amount of pressure to acupoints. There are 9 acupressure points, totaling 27 minutes of stimulation per day. Participants will perform daily acupressure for a total of six weeks.
  In addition all participants will complete a battery of validated questionnaires before, during and after completion of treatment intervention.

SUMMARY:
The goal of this pilot trial is to better understand if acupressure is feasible and tolerable to people with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

- Patient is being treated for Rheumatoid Arthritis (RA) at a Rheumatology Clinic at the University of Michigan or another by rheumatologist and reports being prescribed at least one of the following medications:

* Methotrexate (Trexall, Rheumatrex)
* Hydroxychloroquine (Plaquenil)
* Sulfasalazine (Azulfadine)
* Leflunomide (Arava)
* Tocilizumab (Actemra)
* Tumor necrosis factor inhibitor (TNFi), including:

Adalimumab (Humira) Etanercept (Enbrel) Certolizumab pegol (Cimzia) Golimumab (Simponi) Infliximab (Remicade)

* Abatacept (Orencia)
* Tocilizumab (Actemra)
* Janus kinase inhibitor (JAKi), including:

Tofacitinib (Xeljanz) Baracitinib (Olumiant) Upadacitinib (Rinvoq)

o Rituximab (Rituxan)

Exclusion Criteria:

* Visual or hearing difficulties that would preclude participation,
* Do not speak or read English
* Do not have access to smart phone with access to mobile applications
* Severe psychiatric disorders including history of substance abuse disorders,
* Individuals on high doses of opioids (over 100 oral morphine equivalents)
* Taking blood thinners, including warfarin (Coumadin), dabigatran (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), edoxaban (Savaysa), or betrixaban (Bevyxxa)
* Thrombocytopenia (low platelet count)
* Expecting to receive surgery within the next year for their RA
* Pregnancy or breast feeding, or anticipate pregnancy in next year,
* Actively applying for disability or compensation, or actively involved in litigation.
* Anything at the discretion of the principal investigator or study team

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Murphy, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupressure: The self-acupressure intervention was delivered using the modified MeTime Acupressure mobile application (App) in addition to in-person or virtual instruction via study staff.
  Acupressure: The MeTime Acupressure app was loaded onto computer tablets or smart phones by the participants. Participants also received an AcuWand to be used in association with the acupressure app to help participants apply the correct amount of pressure to acupoints. There were 9 acupressure points, totaling 27 minutes of stimulation per day. Participants performed daily acupressure for a total of six weeks.
  In addition all participants completed a battery of validated questionnaires before, during, and after completion of treatment intervention.
Period: Overall Study
Arm/Group | Acupressure
Started | 14
Day 42 - End of Treatment | 6
Completed | 4
Not Completed | 10
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Acupressure
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Self-performed Acupressure in Patients With Rheumatoid Arthritis Assessed by the Number of Sessions Completed
Description: Feasibility of self-performed acupressure in patients with rheumatoid arthritis assessed by the number of study sessions completed by participants. Results reflect the number of participants who responded to all of the surveys administered at the Day 42 visit.
Time Frame: up to day 42 (during acupressure)
Measure: Count of Participants; unit: Participants
Arm/Group | Acupressure
Number analyzed (Participants) | 14
Participants | 6

2. Primary Outcome: Acceptability of Self-performed Acupressure in Patients With RA Assessed by Acupressure Tolerability Scale at Day 42 - Question 1
Description: The Acupressure Tolerability Scale was comprised of 4 questions for participants to complete. Each question used a different scoring method, so the questions are reported as separate outcomes.
  Question 1 asked whether participants were able to perform acupressure for the required time each day. Responses were on a 0-10 scale with 0 being 'not at all' and 10 being 'all of the time.'
Time Frame: Day 42 (during acupressure)
Population: Only participants who completed the survey at the Day 42 session were analyzed. Neither a p-value nor an estimation parameter were used due to the small participant sample size.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 6
score on a scale | 7 [3 to 10]

3. Primary Outcome: Acceptability of Self-performed Acupressure in Patients With RA Assessed by Acupressure Tolerability Scale at Day 42 - Question 2
Description: The Acupressure Tolerability Scale was comprised of 4 questions for participants to complete. Each question used a different scoring method, so the questions are reported as separate outcomes.
  Question 2 asked whether participants had to stop performing acupressure at any point during administration. Responses were on a 0-10 scale with 0 being 'not at all' and 10 being 'all of the time.'
Time Frame: Day 42 (during acupressure)
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 6
score on a scale | 4 [1 to 8]

4. Primary Outcome: Acceptability of Self-performed Acupressure in Patients With RA Assessed by Acupressure Tolerability Scale at Day 42 - Question 3
Description: The Acupressure Tolerability Scale was comprised of 4 questions for participants to complete. Each question used a different scoring method, so the questions are reported as separate outcomes.
  Question 3 asked whether participants stopped acupressure because of pain in the hands. Responses could either be Yes or No. The results represent the number of participants who responded 'Yes' to this question.
Time Frame: Day 42 (during acupressure)
Population: Only participants who completed the survey at the Day 42 session were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupressure
Number analyzed (Participants) | 6
Participants | 2

5. Primary Outcome: Acceptability of Self-performed Acupressure in Patients With RA Assessed by Acupressure Tolerability Scale at Day 42 - Question 4
Description: The Acupressure Tolerability Scale was comprised of 4 questions for participants to complete. Each question used a different scoring method, so the questions are reported as separate outcomes.
  Question 4 asked whether participants stopped acupressure because of pain at the acupoint, i.e., the place on the body where pressure was being applied. Responses could either be Yes or No. The results represent the number of participants who responded 'Yes' to this question.
Time Frame: Day 42 (during acupressure)
Population: Only participants who completed the survey at the Day 42 session were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupressure
Number analyzed (Participants) | 6
Participants | 1

6. Secondary Outcome: Change in Fibromyalgia Survey Questionnaire
Description: The fibromyalgia survey questionnaire comprises a measure of widespread body pain (0-19 points; one point per body location) and an assessment of comorbid symptoms (0-12 points including fatigue/depression/sleep/cognition) which are added together for a total possible score of 0-31 (0 being the lowest score, reflecting the least amount of pain and co-morbid symptoms; 31 being the highest score, reflecting the highest amount of pain and co-morbid symptoms captured on the scale). Scores are reported as a single composite score of the total number of points. A score of 13 or higher is needed for the Fibromyalgia diagnosis. This can arise from multiple combinations of the widespread pain and symptom severity scores. Results are an average of the participants' scores collected at baseline and at Day 42.
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session. Neither a p-value nor an estimation parameter were used due to the small participant sample size.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 10.8 [3 to 19.5]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 7.6 [2 to 23.8]

7. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Physical Functioning
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function and pain intensity. This physical function subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lowest/worst physical functioning) and 20 (reflecting highest/best physical functioning).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 15.6 [9 to 20]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 16.3 [8 to 20]

8. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Anxiety
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function, and pain intensity. This anxiety subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lowest anxiety) and 20 (reflecting highest anxiety).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 7.8 [4 to 12]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 6 [4 to 10]

9. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Depression
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function and pain intensity. This depression subscale consists of 3 questions, which can result in a raw score of between 3 (reflecting lowest depression) and 15 (reflecting highest depression).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 6.9 [4 to 14]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 5.5 [4 to 11]

10. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Fatigue
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function, and pain intensity. This fatigue subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lowest fatigue) and 20 (reflecting highest fatigue).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 10.9 [4 to 20]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 8.2 [4 to 18]

11. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Sleep Disturbance
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function, and pain intensity. This sleep subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lower sleep disturbance and therefore better sleep quality) and 20 (reflecting highest sleep disturbance and therefore worse sleep quality).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 10.8 [9 to 14]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 11.2 [10 to 14]

12. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Social Participation
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function, and pain intensity. This social participation subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lowest/worst ability to participate in social roles and activities) and 20 (reflecting highest/best ability to participate in social roles and activities).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 13.5 [9 to 16]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 13.7 [6 to 16]

13. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Pain Interference
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function, and pain intensity. This pain interference subscale consists of 4 questions, which can result in a raw score of between 4 (reflecting lowest pain interference) and 20 (reflecting highest pain interference).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 10.5 [4 to 18]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 8.7 [4 to 20]

14. Secondary Outcome: Change in the Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS-29 +2) - Cognitive Function
Description: The PROMIS-29 plus 2 Profile v2.1 is designed for adults ≥18 years of age and includes 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function. This cognitive function subscale consists of 2 questions, which can result in a raw score of between 2 (reflecting lowest/worst cognitive function) and 10 (reflecting highest/best cognitive function).
Time Frame: Baseline to Day 42
Population: 14 participants completed the survey at baseline. Only 6 participants completed the survey at the Day 42 session.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acupressure
Number analyzed (Participants) | 14
score on a scale
  Baseline | 8 [5 to 10]
  Day 42: number analyzed (Participants) | 6
  Day 42 | 8.2 [6 to 10]

ADVERSE EVENTS:
Time Frame: 63 days
Arm/Group | Acupressure
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupressure (N=14)
Hip pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT05412121/Prot_SAP_000.pdf